CLINICAL TRIAL: NCT03740048
Title: A Randomized Pilot Study of Hemodialysis Initiation Comparing Twice-Weekly Hemodialysis Plus Dialysis-Sparing Therapy Versus Thrice-Weekly Hemodialysis (The TWOPLUS-HD Trial)
Brief Title: A Pilot Trial of Twice-weekly Versus Thrice-weekly Hemodialysis in Patients With Incident End-stage Kidney Disease
Acronym: TWOPLUS-HD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00054726
Record Dates: First submitted 2018-11-09; First posted 2018-11-14 (Actual); Results first posted 2023-06-05 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2022-04

CONDITIONS: End Stage Renal Failure on Dialysis
Keywords: Hemodialysis; Kidney Disease; Kidney Function
MeSH Terms: conditions — Kidney Diseases | interventions — Renal Dialysis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hemodialysis and Pharmacologic Therapy (Experimental): Hemodialysis regimen at the initiation of dialysis treatment: Twice-weekly hemodialysis plus adjunctive pharmacologic therapy (loop diuretic, potassium-binding agent, and sodium bicarbonate) for six consecutive weeks, continued by thrice-weekly hemodialysis (intervention group)
  Interventions: Other: Hemodialysis; Drug: Patiromer Oral Product
- Conventional Hemodialysis Regimen (Active Comparator): Hemodialysis regimen at the initiation of dialysis treatment: thrice-weekly hemodialysis
  Interventions: Other: Hemodialysis

INTERVENTIONS:
Other: Hemodialysis — Hemodialysis frequency will differ in the first six weeks of hemodialysis therapy between the two treatment arms.
Drug: Patiromer Oral Product — Participants in the intervention group who develop hyperkalemia, during the first six weeks of receiving hemodialysis twice per week, will be treated with Patiromer.
  Arms: Hemodialysis and Pharmacologic Therapy

SUMMARY:
The optimal frequency of hemodialysis treatments in patients with incident end-stage kidney disease in not known. This pilot trial will randomize patients with incident end-stage kidney disease due to chronic kidney disease progression to two different regimens of hemodialysis: i) twice-weekly hemodialysis for six weeks with adjuvant pharmacologic medications followed by thrice-weekly hemodialysis, or ii) thrice-weekly hemodialysis. The study will test feasibility of stepwise hemodialysis, and the effects of the two regimens of hemodialysis on residual kidney function.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Incident ESKD from CKD progression (including a failing renal transplant)
* Are deemed to require dialysis initiation by the treating nephrologist
* Have elected HD for renal replacement therapy (RRT)

Exclusion Criteria:

* Have urine output <500ml per day
* Have ESKD as a result of severe acute kidney injury (AKI) (stage 3 AKI defined by Acute Kidney Injury Network [AKIN]) criteria)
* Abrupt decline in kidney function preceding HD therapy initiation (i.e., if eGFR was ≥30 mL/min/1.73 m2 3 months prior to the initiation of dialysis therapy)
* Are scheduled to undergo transplantation from a live donor within the next 6 months
* Have an active diagnosis of hepatorenal syndrome
* Have a significant malignancy that is likely to impact survival
* Have a medical condition that would jeopardize the safety of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Murea, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
After study completion, de-identified participant data may be provided to other researchers in the filed if requested. The request(s) will be reviewed by the principal investigator and other study members to determine if appropriate.
Supporting Information: Study Protocol, SAP
Time Frame: 2-4 months

REFERENCES:
- [Background] National Kidney Foundation. KDOQI Clinical Practice Guideline for Hemodialysis Adequacy: 2015 update. Am J Kidney Dis. 2015 Nov;66(5):884-930. doi: 10.1053/j.ajkd.2015.07.015. PMID 26498416
- [Background] Lowrie EG, Laird NM, Parker TF, Sargent JA. Effect of the hemodialysis prescription on patient morbidity: report from the National Cooperative Dialysis Study. N Engl J Med. 1981 Nov 12;305(20):1176-81. doi: 10.1056/NEJM198111123052003. PMID 7027040
- [Background] Eknoyan G, Beck GJ, Cheung AK, Daugirdas JT, Greene T, Kusek JW, Allon M, Bailey J, Delmez JA, Depner TA, Dwyer JT, Levey AS, Levin NW, Milford E, Ornt DB, Rocco MV, Schulman G, Schwab SJ, Teehan BP, Toto R; Hemodialysis (HEMO) Study Group. Effect of dialysis dose and membrane flux in maintenance hemodialysis. N Engl J Med. 2002 Dec 19;347(25):2010-9. doi: 10.1056/NEJMoa021583. PMID 12490682
- [Background] Paniagua R, Amato D, Vonesh E, Correa-Rotter R, Ramos A, Moran J, Mujais S. Effects of increased peritoneal clearances on mortality rates in peritoneal dialysis: ADEMEX, a prospective, randomized, controlled trial. J Am Soc Nephrol. 2002 May;13(5):1307-1320. doi: 10.1681/ASN.V1351307. PMID 11961019
- [Background] Lo WK, Ho YW, Li CS, Wong KS, Chan TM, Yu AW, Ng FS, Cheng IK. Effect of Kt/V on survival and clinical outcome in CAPD patients in a randomized prospective study. Kidney Int. 2003 Aug;64(2):649-56. doi: 10.1046/j.1523-1755.2003.00098.x. PMID 12846762
- [Background] Li Y, Jin Y, Kapke A, Pearson J, Saran R, Port FK, Robinson BM. Explaining trends and variation in timing of dialysis initiation in the United States. Medicine (Baltimore). 2017 May;96(20):e6911. doi: 10.1097/MD.0000000000006911. PMID 28514305
- [Background] Chin AI, Appasamy S, Carey RJ, Madan N. Feasibility of Incremental 2-Times Weekly Hemodialysis in Incident Patients With Residual Kidney Function. Kidney Int Rep. 2017 Jun 21;2(5):933-942. doi: 10.1016/j.ekir.2017.06.005. eCollection 2017 Sep. PMID 29270499
- [Background] Lin YF, Huang JW, Wu MS, Chu TS, Lin SL, Chen YM, Tsai TJ, Wu KD. Comparison of residual renal function in patients undergoing twice-weekly versus three-times-weekly haemodialysis. Nephrology (Carlton). 2009 Feb;14(1):59-64. doi: 10.1111/j.1440-1797.2008.01016.x. Epub 2008 Nov 19. PMID 19019171
- [Background] Zhang M, Wang M, Li H, Yu P, Yuan L, Hao C, Chen J, Kalantar-Zadeh K. Association of initial twice-weekly hemodialysis treatment with preservation of residual kidney function in ESRD patients. Am J Nephrol. 2014;40(2):140-50. doi: 10.1159/000365819. Epub 2014 Aug 23. PMID 25171342
- [Background] Shafi T, Jaar BG, Plantinga LC, Fink NE, Sadler JH, Parekh RS, Powe NR, Coresh J. Association of residual urine output with mortality, quality of life, and inflammation in incident hemodialysis patients: the Choices for Healthy Outcomes in Caring for End-Stage Renal Disease (CHOICE) Study. Am J Kidney Dis. 2010 Aug;56(2):348-58. doi: 10.1053/j.ajkd.2010.03.020. Epub 2010 Jun 3. PMID 20605303
- [Background] Termorshuizen F, Dekker FW, van Manen JG, Korevaar JC, Boeschoten EW, Krediet RT; NECOSAD Study Group. Relative contribution of residual renal function and different measures of adequacy to survival in hemodialysis patients: an analysis of the Netherlands Cooperative Study on the Adequacy of Dialysis (NECOSAD)-2. J Am Soc Nephrol. 2004 Apr;15(4):1061-70. doi: 10.1097/01.asn.0000117976.29592.93. PMID 15034110
- [Background] Marquez IO, Tambra S, Luo FY, Li Y, Plummer NS, Hostetter TH, Meyer TW. Contribution of residual function to removal of protein-bound solutes in hemodialysis. Clin J Am Soc Nephrol. 2011 Feb;6(2):290-6. doi: 10.2215/CJN.06100710. Epub 2010 Oct 28. PMID 21030575
- [Background] Weir MR, Bakris GL, Bushinsky DA, Mayo MR, Garza D, Stasiv Y, Wittes J, Christ-Schmidt H, Berman L, Pitt B; OPAL-HK Investigators. Patiromer in patients with kidney disease and hyperkalemia receiving RAAS inhibitors. N Engl J Med. 2015 Jan 15;372(3):211-21. doi: 10.1056/NEJMoa1410853. Epub 2014 Nov 21. PMID 25415805
- [Background] Bakris GL, Pitt B, Weir MR, Freeman MW, Mayo MR, Garza D, Stasiv Y, Zawadzki R, Berman L, Bushinsky DA; AMETHYST-DN Investigators. Effect of Patiromer on Serum Potassium Level in Patients With Hyperkalemia and Diabetic Kidney Disease: The AMETHYST-DN Randomized Clinical Trial. JAMA. 2015 Jul 14;314(2):151-61. doi: 10.1001/jama.2015.7446. PMID 26172895
- [Background] Pitt B, Bakris GL, Bushinsky DA, Garza D, Mayo MR, Stasiv Y, Christ-Schmidt H, Berman L, Weir MR. Effect of patiromer on reducing serum potassium and preventing recurrent hyperkalaemia in patients with heart failure and chronic kidney disease on RAAS inhibitors. Eur J Heart Fail. 2015 Oct;17(10):1057-65. doi: 10.1002/ejhf.402. Epub 2015 Oct 12. PMID 26459796
- [Background] Kovesdy CP, Regidor DL, Mehrotra R, Jing J, McAllister CJ, Greenland S, Kopple JD, Kalantar-Zadeh K. Serum and dialysate potassium concentrations and survival in hemodialysis patients. Clin J Am Soc Nephrol. 2007 Sep;2(5):999-1007. doi: 10.2215/CJN.04451206. Epub 2007 Aug 16. PMID 17702709
- [Background] Wu DY, Shinaberger CS, Regidor DL, McAllister CJ, Kopple JD, Kalantar-Zadeh K. Association between serum bicarbonate and death in hemodialysis patients: is it better to be acidotic or alkalotic? Clin J Am Soc Nephrol. 2006 Jan;1(1):70-8. doi: 10.2215/CJN.00010505. Epub 2005 Nov 23. PMID 17699193
- [Background] Daugirdas JT. Estimating Time-averaged Serum Urea Nitrogen Concentration during Various Urine Collection Periods: A Prediction Equation for Thrice Weekly and Biweekly Dialysis Schedules. Semin Dial. 2016 Nov;29(6):507-509. doi: 10.1111/sdi.12554. Epub 2016 Oct 4. PMID 27699876
- [Background] Daugirdas JT, Depner TA, Greene T, Levin NW, Chertow GM, Rocco MV; Frequent Hemodialysis Network Trial Group. Standard Kt/Vurea: a method of calculation that includes effects of fluid removal and residual kidney clearance. Kidney Int. 2010 Apr;77(7):637-44. doi: 10.1038/ki.2009.525. Epub 2010 Jan 27. PMID 20107428
- [Background] Jansen MA, Hart AA, Korevaar JC, Dekker FW, Boeschoten EW, Krediet RT; NECOSAD Study Group. Predictors of the rate of decline of residual renal function in incident dialysis patients. Kidney Int. 2002 Sep;62(3):1046-53. doi: 10.1046/j.1523-1755.2002.00505.x. PMID 12164889
- [Derived] Murea M, Highland BR, Yang W, Dressler E, Russell GB. Patient-reported outcomes in a pilot clinical trial of twice-weekly hemodialysis start with adjuvant pharmacotherapy and transition to thrice-weekly hemodialysis vs conventional hemodialysis. BMC Nephrol. 2022 Sep 27;23(1):322. doi: 10.1186/s12882-022-02946-w. PMID 36167537
- [Derived] Murea M, Patel A, Highland BR, Yang W, Fletcher AJ, Kalantar-Zadeh K, Dressler E, Russell GB. Twice-Weekly Hemodialysis With Adjuvant Pharmacotherapy and Transition to Thrice-Weekly Hemodialysis: A Pilot Study. Am J Kidney Dis. 2022 Aug;80(2):227-240.e1. doi: 10.1053/j.ajkd.2021.12.001. Epub 2021 Dec 18. PMID 34933066
- [Derived] Murea M, Moossavi S, Fletcher AJ, Jones DN, Sheikh HI, Russell G, Kalantar-Zadeh K. Renal replacement treatment initiation with twice-weekly versus thrice-weekly haemodialysis in patients with incident dialysis-dependent kidney disease: rationale and design of the TWOPLUS pilot clinical trial. BMJ Open. 2021 May 24;11(5):e047596. doi: 10.1136/bmjopen-2020-047596. PMID 34031117
- [Derived] Murea M. Precision medicine approach to dialysis including incremental and decremental dialysis regimens. Curr Opin Nephrol Hypertens. 2021 Jan;30(1):85-92. doi: 10.1097/MNH.0000000000000667. PMID 33165001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 51 patients consented to participate and enrolled for the study. 48 patients were randomized to treatment with twice-weekly HD and adjuvant pharmacotherapy for 6 weeks followed by thrice-weekly HD (n = 23) or continued usual care treatment with thrice-weekly HD (n = 25).
Pre-assignment Details: 77 patients (41%) were approached for study participation. Of those, 51 (66%) consented to participate, resulting in 48 patients randomized to treatment with twice-weekly HD and adjuvant pharmacotherapy for 6 weeks followed by thrice-weekly HD (n = 23) or continued usual care treatment with thrice-weekly HD (n = 25).
Period: Overall Study
Arm/Group | Hemodialysis and Pharmacologic Therapy | Conventional Hemodialysis Regimen
Started | 23 | 25
Completed | 17 | 16
Not Completed | 6 | 9
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Death | 1 | 6
Not completed — Switched to thrice-weekly HD | 2 | 0
Not completed — Switched to Peritoneal Dialysis | 2 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Non-compliance with HD | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hemodialysis and Pharmacologic Therapy | Conventional Hemodialysis Regimen | Total
Number analyzed (Participants) | 23 | 25 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (15.0) | 63.3 (12.8) | 61.3 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 13 | 14 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 16 | 27
  White | 11 | 8 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 32.5 (9.4) | 31.8 (8.4) | 32.1 (8.8)
Body surface area [Mean (Standard Deviation); unit: m^2] | 2.1 (0.2) | 2.0 (0.3) | 2.06 (0.3)

OUTCOME MEASURES:

1. Primary Outcome: Patients' Adherence to Study Protocol
Description: ≥95% of participants randomized in the intervention group will adhere to the HD regimen. All participants who completed 6 and 12 months of follow-up completed interdialytic timed urine collections - Patient adherence to the study protocol was assessed by the number of participants randomized to each intervention who adhered to the study protocol and at 6 months and at 12 months
Time Frame: 6 months, 12 months, 24 months
Population: Participants were censored at death, HD withdrawal, or conversion to peritoneal dialysis. Not included in data analysis were participants who withdrew consent, were withdrawn from the study because of nonadherence to HD treatments, or were lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Hemodialysis and Pharmacologic Therapy | Conventional Hemodialysis Regimen
Number analyzed (Participants) | 23 | 25
Participants
  Patients adherence to study protocol | 22 | 24
  interdialytic timed urine collections at 6 month followup: number analyzed (Participants) | 19 | 19
  interdialytic timed urine collections at 6 month followup | 19 | 19
  interdialytic timed urine collections at 12 month followup: number analyzed (Participants) | 10 | 10
  interdialytic timed urine collections at 12 month followup | 10 | 10

2. Secondary Outcome: 24-hour Urine Volume
Description: Residual renal clearance was calculated based on 24-hour urine collection performed at baseline at enrollment; and interdialytic urine collection performed at baseline, 6 Weeks, 12 Weeks and 24 Weeks
Time Frame: Baseline, 6 Weeks, 12 Weeks, 24 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/day
Arm/Group | Hemodialysis and Pharmacologic Therapy | Conventional Hemodialysis Regimen
Number analyzed (Participants) | 23 | 25
mL/day
  Urine volume at Baseline | 914 [654 to 1174] | 1424 [976 to 1872]
  Urine volume at Week 6: number analyzed (Participants) | 19 | 17
  Urine volume at Week 6 | 504 [335 to 673] | 553 [384 to 723]
  Urine volume at 12 weeks: number analyzed (Participants) | 19 | 19
  Urine volume at 12 weeks | 479 [288 to 670] | 484 [292 to 676]
  Urine volume at 24 Weeks: number analyzed (Participants) | 17 | 15
  Urine volume at 24 Weeks | 862 [624 to 1099] | 876 [638 to 1114]

3. Secondary Outcome: Change in Residual Kidney Function - Urea Clearance
Description: Residual renal clearance was calculated based on 24-hour urine collection performed at baseline at enrollment; and interdialytic urine collection performed during weeks 6, 12, and 24.
Time Frame: Baseline, 6 Weeks, 12 Weeks, 24 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min/1.73m^2
Arm/Group | Hemodialysis and Pharmacologic Therapy | Conventional Hemodialysis Regimen
Number analyzed (Participants) | 23 | 25
mL/min/1.73m^2
  Baseline Renal Urea Clearance: number analyzed (Participants) | 18 | 17
  Baseline Renal Urea Clearance | 3.3 [2.0 to 4.5] | 4.1 [2.9 to 5.3]
  Week 6 Renal Urea Clearance: number analyzed (Participants) | 19 | 17
  Week 6 Renal Urea Clearance | 2.3 [1.6 to 2.9] | 2.3 [1.6 to 3.0]
  Week 12 Renal Urea Clearance: number analyzed (Participants) | 19 | 19
  Week 12 Renal Urea Clearance | 2.1 [1.4 to 2.8] | 2.0 [1.4 to 2.7]
  Week 24 Renal Urea Clearance: number analyzed (Participants) | 17 | 15
  Week 24 Renal Urea Clearance | 1.6 [0.9 to 2.2] | 2.2 [1.6 to 2.8]

4. Secondary Outcome: Change in Residual Kidney Function - Creatinine Clearance
Description: as for outcome 3
Time Frame: Baseline, 6 Weeks, 12 Weeks, 24 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min/1.73m^2
Arm/Group | Hemodialysis and Pharmacologic Therapy | Conventional Hemodialysis Regimen
Number analyzed (Participants) | 23 | 25
mL/min/1.73m^2
  Baseline Renal Creatinine Clearance: number analyzed (Participants) | 18 | 18
  Baseline Renal Creatinine Clearance | 8.4 [5.6 to 11.3] | 10.8 [8.1 to 13.5]
  Week 6 Renal Creatinine Clearance: number analyzed (Participants) | 15 | 19
  Week 6 Renal Creatinine Clearance | 5.5 [2.9 to 8.1] | 6.8 [4.7 to 9.0]
  Week 12 Renal Creatinine Clearance: number analyzed (Participants) | 15 | 17
  Week 12 Renal Creatinine Clearance | 5.3 [3.2 to 7.4] | 5.8 [4.1 to 7.5]
  Week 24 Renal Creatinine Clearance: number analyzed (Participants) | 16 | 15
  Week 24 Renal Creatinine Clearance | 5.6 [3.9 to 7.3] | 5.4 [3.7 to 7.2]

ADVERSE EVENTS:
Time Frame: Monthly basis up to Year 2
Description: Three patients from the conventional group were excluded from the analysis due to insufficient data resulting from early consent withdrawal, non-compliance with HD due to no-show, and loss to follow-up. In addition, one patient from the incremental group was also not included in the analysis due to consent withdrawal.
Arm/Group | Hemodialysis and Pharmacologic Therapy | Conventional Hemodialysis Regimen
All-Cause Mortality (participants affected / at risk) | 1/22 | 6/22
Serious Adverse Events (participants affected / at risk) | 11/22 | 12/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hemodialysis and Pharmacologic Therapy (N=22) | Conventional Hemodialysis Regimen (N=22)
hospitalization (Cardiac disorders) | 1 | 4 — Cardiovascular
Hospitalization (Vascular disorders) | 4 | 1 — Cerebrovascular
hospitalization (General disorders) | 0 | 6 — Fluid manageme
hospitalization (General disorders) | 1 | 0 — Hyperkalemia
hospitalization (Nervous system disorders) | 0 | 5 — Encephalopathy
hospitalization (Infections and infestations) | 2 | 0 — Vascular access infection
hospitalization (General disorders) | 0 | 1 — Vascular access complication, noninfectious
hospitalization (Infections and infestations) | 4 | 9 — Infection, not related to vascular access
hospitalization (General disorders) | 6 | 7 — other

LIMITATIONS AND CAVEATS:
Our results should be interpreted in the context of several limitations. Given (1) the imbalances in baseline characteristics between the 2 groups, (2) the small sample size, and (3) the time-delineated twice-weekly HD, the effect estimates are solely exploratory. Our testing of a time-delineated prescription of twice-weekly HD for 6 weeks may leave lingering concerns as to whether incremental HD with longer periods of twice-weekly HD can be effectively and safely implemented.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/48/NCT03740048/Prot_SAP_001.pdf
  • Informed Consent Form (2021-05-07): https://cdn.clinicaltrials.gov/large-docs/48/NCT03740048/ICF_002.pdf